CLINICAL TRIAL: NCT04820686
Title: A Randomized Phase 2a, Multicenter, Open-Label, Multiple-Cohort Study Evaluating Regimens Containing Vebicorvir in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Study Evaluating Treatment Regimens Containing Vebicorvir (ABI-H0731) in Participants With Chronic Hepatitis B Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Assembly Biosciences (Industry)
Collaborators: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-H0731-204
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Chronic Hepatitis B
Keywords: cHBV; HBV; hepatitis B; vebicorvir; VBR; AB-729
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VBR + AB-729 + SOC NrtI (Experimental): Participants with cHBV received VBR + AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up.
  Interventions: Drug: VBR; Drug: AB-729; Drug: SOC NrtI
- VBR + SOC NrtI (Other): Participants with cHBV received VBR + SOC NrtI for 48 weeks followed by 48 weeks in follow-up. This treatment was used as a reference regimen.
  Interventions: Drug: VBR; Drug: SOC NrtI
- AB-729 + SOC NrtI (Other): Participants with cHBV received AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up. This treatment was used as a reference regimen.
  Interventions: Drug: AB-729; Drug: SOC NrtI

INTERVENTIONS:
Drug: VBR — VBR is an HBV core protein inhibitor. Participants will receive VBR 300 mg tablets orally once daily (QD).
  Other Names: Vebicorvir, ABI-H0731
  Arms: VBR + AB-729 + SOC NrtI; VBR + SOC NrtI
Drug: AB-729 — AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants will receive a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  Arms: AB-729 + SOC NrtI; VBR + AB-729 + SOC NrtI
Drug: SOC NrtI — Participants will receive their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
  Other Names: Entecavir (ETV); Tenofovir disoproxil fumarate (TDF); Tenofovir alafenamide (TAF)

SUMMARY:
The purpose of this study is to determine if vebicorvir (VBR, ABI-H0731) in combination with AB-729 is safe and effective in participants with chronic hepatitis B infection (cHBV) receiving a standard of care nucleos(t)ide/reverse transcriptase inhibitor (SOC NrtI).

DETAILED DESCRIPTION:
The initial cohort of participants will be enrolled in 3 treatment groups receiving 1) VBR + AB-729 + SOC NrtI, 2) VBR + SOC NrtI, or 3) AB-729 + SOC NrtI for up to 48 weeks. At Week 48, all participants will have an assessment of Treatment Stopping Criteria. Any participant who meets the Treatment Stopping Criteria, will discontinue their assigned treatment including NrtI and will remain in follow-up through Week 96. The participants who do not meet the Treatment Stopping Criteria will continue treatment with NrtI alone and will remain in follow-up through Week 96. Up to an additional 2 cohorts may be added to the study in future protocol amendments.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 36 kg/m^2 and a minimum body weight of 45 kg (inclusive)
* Female participants must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day 1
* Chronic Hepatitis B defined as HBV infection documented for ≥6 months prior to Screening
* Hepatitis B 'e' antigen (HBeAg) negative at least 3 months prior to Screening Visit (historical documentation) AND at the Screening Visit
* Virologically suppressed on SOC NrtI therapy with nonquantifiable HBV DNA for at least 6 months prior to Screening
* On a stable SOC NrtI regimen of ETV, TDF, or TAF for >12 months
* HBsAg ≥100 international units/mL at Screening
* Lack of bridging fibrosis or cirrhosis
* Agreement to comply with protocol-specified contraceptive requirements
* In good general health, except for cHBV, in the opinion of the Investigator
* Able to take oral medication and willing to receive subcutaneous injections of AB-729.

Exclusion Criteria:

* Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis D virus (HDV), acute hepatitis A virus (HAV), or acute hepatitis E virus (HEV)
* Females who are lactating or wish to become pregnant during the course of the study
* History of liver transplant or evidence of advanced liver disease, cirrhosis, or hepatic decompensation at any time prior to, or at the time of Screening
* History of persistent alcohol abuse or illicit drug abuse within 3 years prior to Screening
* Clinically significant diseases or conditions, such as cardiac disease, including poorly-controlled or unstable hypertension; pulmonary disease; chronic or recurrent renal or urinary tract disease; liver disease other than cHBV; endocrine disorder; autoimmune disorder; poorly controlled diabetes mellitus; neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment; ongoing infection or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that, in the opinion of the Investigator or the Sponsor, makes the subject unsuitable for study participation
* History of hepatocellular carcinoma (HCC)
* History of malignancy other than HCC unless the subject's malignancy has been in complete remission off chemotherapy and without additional medical or surgical interventions during the 3 years before Screening
* History or presence at Screening of electrocardiogram (ECG) abnormalities deemed clinically significant, in the opinion of the Investigator
* History of hypersensitivity or idiosyncratic reaction to any components or excipients of the investigational drugs
* History of any significant food or drug-related allergic reactions such as anaphylaxis or Stevens-Johnson syndrome
* Exclusionary laboratory results at Screening:

  1. Platelet count <100,000/mm^3
  2. Albumin <3 g/dL
  3. Direct bilirubin >1.2× upper limit of normal (ULN)
  4. ALT ≥5× ULN
  5. Serum alpha fetoprotein (AFP) ≥100 ng/mL. If AFP at Screening is > ULN but <100 ng/mL, the subject is eligible if hepatic imaging prior to initiation of study drug reveals no lesions indicative of possible HCC
  6. International Normalized Ratio (INR) >1.5× ULN
  7. Estimated creatinine clearance (CrCl) <50 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight at Screening
  8. Any other laboratory abnormality deemed clinically significant by the Investigator
* Current or prior use of prohibited (per protocol) concomitant medications from 28 days prior to Day 1.
* Current or prior treatment for cHBV with:

  * Lamivudine, telbivudine or adefovir (any duration)
  * HBV core inhibitor (any duration)
  * siRNA or other oligonucleotide therapeutic (any duration)
  * Interferon in the 6 months prior to Screening
  * Any investigational agent for cHBV in the 6 months prior to Screening.
* Participation in another clinical study of a drug or device whereby the last investigational drug/device administration is within 60 days or 5 half-lives prior to study start.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Australia (8):
  - Saint Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Saint George Hospital - Australia, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Footscray Hospital, Footscray, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Melbourne Health, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Bulgaria (4):
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia-Grad
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski, Sofia
  - Nov Rehabilitatsionen Tsentar EOOD, Stara Zagora
- Canada (6):
  - Vancouver Infectious Disease Centre, Vancouver, British Columbia
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Centre Hospitalier Université de Québec - Université Laval, Québec
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Wellington Regional Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ligat G, Verrier ER, Nassal M, Baumert TF. Hepatitis B virus-host interactions and novel targets for viral cure. Curr Opin Virol. 2021 Aug;49:41-51. doi: 10.1016/j.coviro.2021.04.009. Epub 2021 May 22. PMID 34029994

RESULTS

PARTICIPANT FLOW:
Groups:
- VBR + AB-729 + SOC NrtI: Participants with cHBV received VBR + AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until the study was early terminated
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  AB-729: AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants received a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
- VBR + SOC NrtI: Participants with cHBV received VBR + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until the study was early terminated. This treatment was used as a reference regimen.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
- AB-729 + SOC NrtI: Participants with cHBV received AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until the study was early terminated. This treatment was used as a reference regimen.
  AB-729: AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants received a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
Period: Overall Study
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Started | 32 | 16 | 17
Completed | 2 | 0 | 0
Not Completed | 30 | 16 | 17
Not completed — Withdrawal by Subject | 5 | 2 | 3
Not completed — Study Termination | 25 | 13 | 14
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- VBR + AB-729 + SOC NrtI: Participants with cHBV received VBR + AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until the study was early terminated.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  AB-729: AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants received a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
- Total: Total of all reporting groups
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI | Total
Number analyzed (Participants) | 32 | 16 | 17 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (6.1) | 41 (6.4) | 42 (5.9) | 41 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 10 | 43
  Male | 12 | 3 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 16 | 17 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 6 | 6 | 22
  Black or African American | 4 | 0 | 1 | 5
  American Indian / Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Asian | 17 | 10 | 10 | 37
  Other | 1 | 0 | 0 | 1
Body Weight [Mean (Standard Deviation); unit: kg] | 73.8 (15.77) | 74.2 (15.38) | 69.2 (12.22) | 72.7 (14.75)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.6 (4.21) | 26.1 (4.67) | 24.1 (3.26) | 25.3 (4.12)
Years positive for HBV [Mean (Standard Deviation); unit: years] | 14.5 (7.75) | 13.1 (11.01) | 15.4 (8.78) | 14.4 (8.80)
HBV Genotype [Count of Participants; unit: Participants] — HBV can be differentiated into genotypes and sub-genotypes via genome sequencing. There can be different clinical outcomes and treatment efficacy related to HBV genotype.
  Participants
    A | 4 | 0 | 2 | 6
    B | 6 | 4 | 3 | 13
    B/C | 2 | 0 | 0 | 2
    C | 5 | 2 | 4 | 11
    C/B | 4 | 1 | 2 | 7
    C/E | 1 | 0 | 0 | 1
    D | 6 | 4 | 4 | 14
    D/B | 1 | 0 | 0 | 1
    E | 1 | 0 | 0 | 1
    Unable to Genotype | 2 | 5 | 2 | 9
NrtI at Baseline [Count of Participants; unit: Participants]
  Tenofovir Alafenamide (TAF) | 6 | 3 | 2 | 11
  Tenofovir disoproxil fumarate (TDF) | 18 | 8 | 13 | 39
  Entecavir (ETV) | 8 | 5 | 2 | 15
Years on current HBV treatment [Mean (Standard Deviation); unit: years] | 6.9 (3.92) | 4.8 (2.67) | 5.9 (3.52) | 6.1 (3.61)
HBV DNA (log10 IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 0.7 (0) | 0.7 (0) | 0.7 (0) | 0.7 (0)
HBV RNA (log10 U/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 1.2 (.88) | 1.1 (.69) | 1.4 (.88) | 1.2 (.83)
HBV TNA Quantitative (Log10 U/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 1.2 (.41) | 1.1 (.32) | 1.2 (.49) | 1.1 (.41)
HBcrAg (Log10 U/mL) [Mean (Standard Deviation); unit: Log10 U/mL] | 3.3 (1.22) | 3.3 (1.43) | 3.2 (.89) | 3.3 (1.19)
HBsAg (Log10 IU/mL) [Mean (Standard Deviation); unit: Log10 IU/mL] | 3.4 (.57) | 3.3 (.62) | 3.3 (.56) | 3.3 (.57)
ALT (U/L) [Mean (Standard Deviation); unit: U/L] | 29 (19.8) | 27 (12.8) | 28 (17.3) | 28 (17.4)
Baseline HBeAb [Count of Participants; unit: Participants]
  Negative | 7 | 2 | 0 | 9
  Positive | 25 | 14 | 17 | 56
Baseline HBsAb [Count of Participants; unit: Participants]
  Negative | 32 | 16 | 17 | 65
  Positive | 0 | 0 | 0 | 0
Fibroscan Result (kPa) [Mean (Standard Deviation); unit: kPa] | 5.2 (1.22) | 5.6 (1.04) | 5.0 (1.13) | 5.3 (1.16)
Metavir Fibrosis Stage [Count of Participants; unit: Participants] — FibroScan is a non-invasive liver elastography test. It measures liver elasticity and the score is recorded as a numerical value measured in kilopascals (kPa). The investigator categorizes the Fibrosis stage based on the FibroScan result. F0 is equivalent to 2-7kPa. F1 is equivalent to 7-11 kPa and F3 is equivalent to 11-19kPa. 19kPa or higher is equivalent to F4. A higher stage corresponds to more advanced liver fibrosis.
  Participants
    F0-F2 | 32 | 16 | 17 | 65
    F3 | 0 | 0 | 0 | 0
    F4 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events (AEs)
Time Frame: AEs were collected from the time of signing the informed consent until the final follow-up visit, up to 96 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- VBR + AB-729 + SOC NrtI: Participants with cHBV received VBR + AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until study was early terminated.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  AB-729: AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants received a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
- VBR + SOC NrtI: Participants with cHBV received VBR + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until study was early terminated. This treatment was used as a reference regimen.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 32 | 16 | 17
Participants | 26 | 12 | 12

2. Primary Outcome: Number of Participants With Premature Treatment Discontinuation Due to AEs
Time Frame: AEs were collected from the time of signing the informed consent until the final follow-up visit, up to 96 weeks.
Population: Subjects in the arm receiving only AB-720 and SOC NrtL were not evaluated for VBR discontinuation. Subjects in the arm reviewing only VBR and SOC NrtI were not evaluated for AB-720 discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 32 | 16 | 17
Participants
  VBR discontinuation due to AE: number analyzed (Participants) | 32 | 16 | 0
  VBR discontinuation due to AE | 3 | 1 |
  AB-729 discontinuation due to AE: number analyzed (Participants) | 32 | 0 | 17
  AB-729 discontinuation due to AE | 1 |  | 0

3. Primary Outcome: Number of Participants With One or More Abnormal Laboratory Result
Time Frame: Laboratory results were collected from the time of signing the informed consent until the study was early terminated, up to 96 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 32 | 16 | 17
Participants | 30 | 16 | 16

4. Secondary Outcome: Change From Baseline in Mean log10 Serum Hepatitis B Surface Antigen (HBsAg) On-Treatment
Description: Subjects remained on their assigned oral agents (ie, VBR+NrtI for Groups 1 and 2; NrtI for Group 3) until Week 48 laboratory results required for Treatment Stopping Criteria assessment were available so there are some results past Week 48.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 56.
Population: The number analyzed differs from the overall number analyzed due to early terminated and/or withdrawn subjects.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- VBR + SOC Nrtl: Participants with cHBV received VBR + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until study was early terminated. This treatment was used as a reference regimen.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC Nrtl | AB-729 + SOC NrtI
Number analyzed (Participants) | 32 | 16 | 17
log10 IU/mL
  Week 2: number analyzed (Participants) | 32 | 15 | 17
  Week 2 | -0.3 (.42) | 0 (0.07) | -0.2 (.26)
  Week 4: number analyzed (Participants) | 30 | 16 | 16
  Week 4 | -.3 (.35) | 0 (0.05) | -0.3 (.39)
  Week 8: number analyzed (Participants) | 29 | 14 | 17
  Week 8 | -0.7 (.62) | 0 (.06) | -0.6 (.42)
  Week 12: number analyzed (Participants) | 29 | 15 | 17
  Week 12 | -1.2 (.65) | 0 (.07) | -1.1 (.5)
  Week 16: number analyzed (Participants) | 29 | 14 | 17
  Week 16 | -1.5 (.56) | 0 (.08) | -1.3 (.53)
  Week 20: number analyzed (Participants) | 27 | 15 | 16
  Week 20 | -1.7 (.55) | 0 (.07) | -1.6 (.53)
  Week 24: number analyzed (Participants) | 27 | 15 | 16
  Week 24 | -1.7 (.52) | 0 (.07) | -1.6 (.42)
  Week 28: number analyzed (Participants) | 25 | 15 | 14
  Week 28 | -1.7 (.54) | 0 (.12) | -1.7 (.49)
  Week 32: number analyzed (Participants) | 27 | 15 | 15
  Week 32 | -1.8 (.5) | 0 (0.1) | -1.7 (.43)
  Week 36: number analyzed (Participants) | 26 | 15 | 15
  Week 36 | -1.9 (.53) | 0 (.11) | -1.9 (.45)
  Week 40: number analyzed (Participants) | 27 | 15 | 15
  Week 40 | -1.8 (.54) | 0 (.11) | -1.8 (.5)
  Week 44: number analyzed (Participants) | 27 | 15 | 15
  Week 44 | -1.9 (.54) | 0 (.11) | -1.9 (.47)
  Week 48: number analyzed (Participants) | 26 | 15 | 10
  Week 48 | -1.9 (.52) | 0 (.12) | -1.9 (.51)
  Week 52: number analyzed (Participants) | 20 | 12 | 0
  Week 52 | -1.8 (.53) | 0 (.09) |
  Week 56: number analyzed (Participants) | 7 | 5 | 0
  Week 56 | -1.5 (.35) | -0.1 (.14) |

5. Secondary Outcome: Number of Participants With Serum HBsAg Below the Lower Limit of Quantitation (<LLOQ)
Time Frame: Pre-specified time points up to 96 weeks
Population: Due to early termination of the study, data was not collected or analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With HBV Deoxyribonucleic Acid (DNA) Not Detected (<5 IU/mL)
Time Frame: Week 48
Population: Due to early termination of the study, data was not collected or analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With HBV Ribonucleic Acid (RNA) <LLOQ
Time Frame: Week 48
Population: Due to early termination of the study, data was not collected or analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Mean log10 HBV RNA On-Treatment
Description: as for outcome 4
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and 56.
Population: The number analyzed differs from the overall number analyzed due to early terminated and/or withdrawn subjects.
Measure: Mean (Standard Deviation); unit: log10 U/mL
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 32 | 16 | 17
log10 U/mL
  Week 2: number analyzed (Participants) | 32 | 15 | 17
  Week 2 | -.6 (.75) | -.2 (.7) | -.4 (.48)
  Week 4: number analyzed (Participants) | 27 | 15 | 16
  Week 4 | -.7 (.76) | 0.2 (.77) | -.6 (.86)
  Week 8: number analyzed (Participants) | 27 | 13 | 17
  Week 8 | -.7 (1.01) | 0 (.59) | -0.5 (.65)
  Week 12: number analyzed (Participants) | 26 | 15 | 17
  Week 12 | -.6 (1.0) | 0 (.55) | -0.7 (.78)
  Week 16: number analyzed (Participants) | 28 | 14 | 15
  Week 16 | -0.6 (.94) | 0 (.58) | -0.8 (.6)
  Week 20: number analyzed (Participants) | 27 | 15 | 15
  Week 20 | -0.7 (1.01) | .1 (.59) | -0.8 (.56)
  Week 24: number analyzed (Participants) | 26 | 15 | 15
  Week 24 | -0.5 (.89) | .2 (.54) | -0.7 (.64)
  Week 28: number analyzed (Participants) | 25 | 15 | 13
  Week 28 | -0.9 (1.0) | .2 (.65) | -0.8 (.59)
  Week 32: number analyzed (Participants) | 27 | 15 | 14
  Week 32 | -0.7 (.89) | .1 (.55) | -0.7 (.68)
  Week 36: number analyzed (Participants) | 26 | 15 | 15
  Week 36 | -0.7 (.88) | .1 (.5) | -0.7 (.78)
  Week 40: number analyzed (Participants) | 26 | 14 | 15
  Week 40 | -0.6 (.88) | .1 (.68) | -0.6 (.57)
  Week 44: number analyzed (Participants) | 27 | 14 | 15
  Week 44 | -0.6 (.87) | 0 (.51) | -0.8 (.69)
  Week 48: number analyzed (Participants) | 26 | 15 | 10
  Week 48 | -0.7 (1.03) | -0.1 (.6) | -0.7 (.46)
  Week 52: number analyzed (Participants) | 18 | 11 | 0
  Week 52 | -0.7 (.89) | -0.1 (.6) |
  Week 56: number analyzed (Participants) | 6 | 5 | 0
  Week 56 | -1.0 (1.37) | .2 (.62) |

9. Secondary Outcome: Change From Baseline in Mean log10 Hepatitis B Core-related Antigen (HBcrAg) On-Treatment
Time Frame: Baseline and Week 48
Population: The number analyzed differs from the overall number analyzed due to early terminated and/or withdrawn subjects.
Measure: Mean (Standard Deviation); unit: log10 U/mL
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 32 | 16 | 17
log10 U/mL | -0.4 (.7) | 0 (.58) | -0.3 (.53)

10. Secondary Outcome: Number of Participants With HBsAg Seroconversion
Time Frame: Week 48
Population: Due to early termination of the study, data was not collected or analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Normal Alanine Aminotransferase (ALT)
Time Frame: Baseline and at pre-specified time points up to 96 weeks
Population: Due to early termination of the study, data was not collected or analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Plasma Levels of VBR
Time Frame: Before dosing at Baseline (Day 1) and at pre-specified time points up to 48 weeks, and at Week 52
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Plasma Levels of AB-729
Time Frame: 2 hours after dosing at pre-specified time points up to 40 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Plasma Levels of SOC NrtI (ETV, TDF, TAF)
Time Frame: Before dosing at Baseline (Day 1) and at pre-specified time points up to 48 weeks
Population: Due to early termination of the study, data was not collected or analyzed for secondary outcomes.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Mean log10 Serum Hepatitis B Surface Antigen (HBsAg) Off-Treatment
Time Frame: Weeks 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92 and 96.
Population: Not all subjects reached Week 96 due to study termination.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Groups:
- VBR + AB-729 + SOC NrtI (Discontinued All); VBR + AB-720 + SOC NrtI (Continued NrtI Only): Participants with cHBV received VBR + AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until study was early terminated.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  AB-729: AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants received a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
- VBR + SOC Nrtl (Discontinued All); VBR + SOC Nrtl (Continued NrtI Only): Participants with cHBV received VBR + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until study was early terminated. This treatment was used as a reference regimen.
  VBR: VBR is an HBV core protein inhibitor. Participants received VBR 300 mg tablets orally once daily (QD).
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
- AB-729 + SOC NrtI (Discontinued All); AB-729 + SOC NrtI (Continued NrtI Only): Participants with cHBV received AB-729 + SOC NrtI for 48 weeks followed by 48 weeks in follow-up or until the study was early terminated. This treatment was used as a reference regimen.
  AB-729: AB-729 is a small interfering ribonucleic acid (siRNA) inhibitor of HBV. Participants received a 60-mg subcutaneous injection of AB-729 once every 8 weeks.
  SOC NrtI: Participants received their SOC NrtI (ETV, TDF or TAF) tablet orally as per approved package insert.
Arm/Group | VBR + AB-729 + SOC NrtI (Discontinued All) | VBR + AB-720 + SOC NrtI (Continued NrtI Only) | VBR + SOC Nrtl (Discontinued All) | VBR + SOC Nrtl (Continued NrtI Only) | AB-729 + SOC NrtI (Discontinued All) | AB-729 + SOC NrtI (Continued NrtI Only)
Number analyzed (Participants) | 12 | 11 | 0 | 12 | 7 | 4
log10 IU/mL
  Off-Treatment Week 4 | -1.9 (.51) | -1.6 (.53) |  | 0 (.09) | -1.8 (.75) | -1.8 (.62)
  Off-Treatment Week 8: number analyzed (Participants) | 9 | 7 | 0 | 7 | 6 | 4
  Off-Treatment Week 8 | -1.9 (.54) | -1.4 (.32) |  | 0 (.08) | -1.8 (.7) | -1.8 (.56)
  Off-Treatment Week 12: number analyzed (Participants) | 6 | 8 | 0 | 6 | 6 | 3
  Off-Treatment Week 12 | -1.8 (.54) | -1.4 (.54) |  | -0.1 (.1) | -1.7 (.62) | -2.0 (.18)
  Off-Treatment Week 16: number analyzed (Participants) | 5 | 6 | 0 | 3 | 5 | 3
  Off-Treatment Week 16 | -1.7 (.24) | -1.5 (.64) |  | -0.1 (.09) | -1.4 (.55) | -1.6 (.62)
  Off-Treatment Week 20: number analyzed (Participants) | 3 | 3 | 0 | 2 | 2 | 3
  Off-Treatment Week 20 | -1.8 (.18) | -1.7 (.85) |  | 0 (.06) | -1.2 (.96) | -2.1 (.28)
  Off-Treatment Week 24: number analyzed (Participants) | 3 | 2 | 0 | 2 | 3 | 1
  Off-Treatment Week 24 | -1.7 (.13) | -2.0 (.78) |  | 0 (.01) | -1.3 (.69) | -2.9 (NA) — Only 1 participant
  Off-Treatment Week 28: number analyzed (Participants) | 2 | 2 | 0 | 1 | 2 | 1
  Off-Treatment Week 28 | -1.8 (.13) | -2.0 (.73) |  | 0 (NA) — Only 1 participant | -1.6 (.06) | -3.0 (NA) — Only 1 participant
  Off-Treatment Week 32: number analyzed (Participants) | 2 | 2 | 0 | 1 | 1 | 1
  Off-Treatment Week 32 | -1.7 (.2) | -1.9 (.72) |  | 0.0 (NA) — Only 1 participant, SD is not applicable. | -1.5 (NA) — Only 1 participant, SD is not applicable. | -3.2 (NA) — Only 1 participant, SD is not applicable.
  Off-Treatment Week 36: number analyzed (Participants) | 2 | 2 | 0 | 1 | 1 | 1
  Off-Treatment Week 36 | -1.6 (.04) | -1.8 (.63) |  | 0 (NA) — Only 1 participant, SD is not applicable. | -1.2 (NA) — Only 1 participant, SD is not applicable. | -3.0 (NA) — Only 1 participant, SD is not applicable.
  Off-Treatment Week 40: number analyzed (Participants) | 0 | 2 | 0 | 0 | 1 | 1
  Off-Treatment Week 40 |  | -1.7 (.68) |  |  | -1.2 (NA) — Only 1 participant, SD is not applicable. | -2.9 (NA) — Only 1 participant, SD is not applicable.
  Off-Treatment Week 44: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 1
  Off-Treatment Week 44 |  | -1.6 (.56) |  |  |  | -2.8 (NA) — Only 1 participant, SD is not applicable.
  Off-Treatment Week 48: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Off-Treatment Week 48 |  | -2.2 (NA) — Only 1 participant, SD is not applicable. |  |  |  |

16. Secondary Outcome: Change From Baseline in Mean log10 HBV RNA Off-Treatment
Time Frame: Weeks 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92 and 96.
Population: Due to study early termination, not all subjects reached week 96.
Measure: Mean (Standard Deviation); unit: log10 U/mL
Arm/Group | VBR + AB-729 + SOC NrtI (Discontinued All) | VBR + AB-720 + SOC NrtI (Continued NrtI Only) | VBR + SOC Nrtl (Discontinued All) | VBR + SOC Nrtl (Continued NrtI Only) | AB-729 + SOC NrtI (Discontinued All) | AB-729 + SOC NrtI (Continued NrtI Only)
Number analyzed (Participants) | 12 | 11 | 0 | 12 | 7 | 4
log10 U/mL
  Off-Treatment Week 4: number analyzed (Participants) | 12 | 11 | 0 | 11 | 7 | 4
  Off-Treatment Week 4 | -0.6 (.83) | -0.8 (1.03) |  | -0.1 (.57) | -1.1 (.61) | -0.9 (1.05)
  Off-Treatment Week 8: number analyzed (Participants) | 10 | 7 | 0 | 8 | 6 | 4
  Off-Treatment Week 8 | -0.5 (.93) | -0.5 (1.02) |  | 0 (.36) | -0.8 (.63) | -0.9 (.56)
  Off-Treatment Week 12: number analyzed (Participants) | 6 | 8 | 0 | 6 | 6 | 3
  Off-Treatment Week 12 | -0.7 (1.11) | -0.6 (1.24) |  | -0.2 (.28) | -0.8 (.66) | -1.0 (.78)
  Off-Treatment Week 16: number analyzed (Participants) | 5 | 6 | 0 | 3 | 5 | 3
  Off-Treatment Week 16 | 0 (1.25) | -0.5 (.55) |  | 0.3 (.31) | -0.8 (.66) | -0.9 (.93)
  Off-Treatment Week 20: number analyzed (Participants) | 3 | 3 | 0 | 2 | 3 | 3
  Off-Treatment Week 20 | .7 (.77) | -0.3 (1.45) |  | -0.2 (.01) | -0.6 (.9) | -0.7 (.65)
  Off-Treatment Week 24: number analyzed (Participants) | 3 | 2 | 0 | 2 | 3 | 1
  Off-Treatment Week 24 | .5 (.41) | -0.4 (1.09) |  | -0.4 (.25) | -0.5 (.2) | 0.7 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 28: number analyzed (Participants) | 2 | 2 | 0 | 1 | 2 | 1
  Off-Treatment Week 28 | 0 (0) | -0.8 (.17) |  | -0.7 (NA) — Only 1 participant, standard deviation is not applicable. | -0.6 (.03) | -0.6 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 32: number analyzed (Participants) | 2 | 2 | 0 | 1 | 1 | 1
  Off-Treatment Week 32 | .2 (.3) | -1.0 (1.26) |  | -0.2 (NA) — Only 1 participant, standard deviation is not applicable. | -0.1 (NA) — Only 1 participant, standard deviation is not applicable. | -0.3 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 36: number analyzed (Participants) | 2 | 2 | 0 | 1 | 1 | 1
  Off-Treatment Week 36 | 0 (0) | -1.0 (.51) |  | 0 (NA) — Only 1 participant, standard deviation is not applicable. | .5 (NA) — Only 1 participant, standard deviation is not applicable. | -0.1 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 40: number analyzed (Participants) | 0 | 2 | 0 | 0 | 1 | 1
  Off-Treatment Week 40 |  | -0.9 (.37) |  |  | -0.4 (NA) — Only 1 participant, standard deviation is not applicable. | -0.6 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 44: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 1
  Off-Treatment Week 44 |  | -1.0 (.39) |  |  |  | .1 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 48: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Off-Treatment Week 48 |  | -1.2 (NA) — Only 1 participant, standard deviation is not applicable. |  |  |  |

17. Secondary Outcome: Change From Baseline in Mean log10 Hepatitis B Core-related Antigen (HBcrAg) Off-Treatment
Time Frame: Weeks 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92 and 96.
Population: Due to study early termination, not all subjects reached week 96.
Measure: Mean (Standard Deviation); unit: log10 U/mL
Arm/Group | VBR + AB-729 + SOC NrtI (Discontinued All) | VBR + AB-720 + SOC NrtI (Continued NrtI Only) | VBR + SOC Nrtl (Discontinued All) | VBR + SOC Nrtl (Continued NrtI Only) | AB-729 + SOC NrtI (Discontinued All) | AB-729 + SOC NrtI (Continued NrtI Only)
Number analyzed (Participants) | 12 | 11 | 0 | 12 | 7 | 4
log10 U/mL
  Off-Treatment Week 12: number analyzed (Participants) | 12 | 10 | 0 | 11 | 6 | 4
  Off-Treatment Week 12 | -0.3 (.46) | -0.5 (.81) |  | .1 (.48) | -0.1 (.18) | -0.6 (.70)
  Off-Treatment Week 24: number analyzed (Participants) | 3 | 3 | 0 | 2 | 3 | 2
  Off-Treatment Week 24 | -0.3 (.17) | -0.2 (.15) |  | .8 (1.13) | -0.2 (.06) | -0.2 (.07)
  Off-Treatment Week 36: number analyzed (Participants) | 2 | 2 | 0 | 1 | 1 | 1
  Off-Treatment Week 36 | -0.3 (.07) | -0.2 (.07) |  | 0 (NA) — Only 1 participant, standard deviation is not applicable. | -0.2 (NA) — Only 1 participant, standard deviation is not applicable. | 0 (NA) — Only 1 participant, standard deviation is not applicable.
  Off-Treatment Week 48: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 1
  Off-Treatment Week 48 |  | -0.1 (.14) |  |  |  | 0 (NA) — Only 1 participant, standard deviation is not applicable.

ADVERSE EVENTS:
Time Frame: Baseline and at pre-specified time points up to 96 weeks
Description: Adverse events were regularly assessed through scheduled investigator assessment and laboratory testing.
Arm/Group | VBR + AB-729 + SOC NrtI | VBR + SOC NrtI | AB-729 + SOC NrtI
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 31/32 | 16/16 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VBR + AB-729 + SOC NrtI (N=32) | VBR + SOC NrtI (N=16) | AB-729 + SOC NrtI (N=17)
Covid-19 Pneumonia (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VBR + AB-729 + SOC NrtI (N=32) | VBR + SOC NrtI (N=16) | AB-729 + SOC NrtI (N=17)
COVID-19 (Infections and infestations) | 6 | 5 | 6
Headache (Nervous system disorders) | 8 | 7 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1 | 3
Fatigue (General disorders) | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 1
Injection Site Pain (General disorders) | 3 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 0

LIMITATIONS AND CAVEATS:
Study ABI-H0731-204 was terminated early by the study Sponsor for strategic reasons to prioritize research and development efforts on finite and curative HBV therapies. As a result, not all subjects completed Week 96 and some outcome measures were impacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT04820686/Prot_SAP_000.pdf